CLINICAL TRIAL: NCT00943878
Title: Effect of Administration of Licensed TIV Vaccine on the Safety and Immunogenicity of an Unadjuvanted Sanofi Pasteur H1N1 Influenza Vaccine in Healthy Adult and Elderly Populations
Brief Title: Sanofi H1N1 + TIV - Adults and Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0039; N01AI80003C
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2010-04

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, vaccine, elderly, TIV
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group 3: H1N1+placebo; H1N1+TIV; placebo (Experimental): 200 subjects (100 ages 18-64 years and 100 aged greater than or equal to 65 years) to receive: Day 0, 15 mcg H1N1 Vaccine + placebo; Day 21, 15 mcg H1N1 Vaccine + trivalent influenza vaccine (TIV); and Day 42, placebo.
  Interventions: Biological: Trivalent inactivated influenza vaccine; Biological: Inactivated H1N1 Vaccine; Drug: Placebo
- Group 1: H1N1+placebo; H1N1+placebo; TIV (Experimental): 200 subjects (100 ages 18-64 years and 100 aged greater than or equal to 65 years) to receive: Day 0, 15 mcg H1N1 Vaccine + placebo; Day 21, 15 mcg H1N1 Vaccine + placebo; and Day 42, trivalent influenza vaccine (TIV).
  Interventions: Biological: Trivalent inactivated influenza vaccine; Biological: Inactivated H1N1 Vaccine; Drug: Placebo
- Group 2: H1N1+TIV; H1N1+placebo; placebo (Experimental): 200 subjects (100 ages 18-64 years and 100 aged greater than or equal to 65 years) to receive: Day 0, 15 mcg H1N1 Vaccine + trivalent influenza vaccine (TIV); Day 21, 15 mcg H1N1 Vaccine + placebo; and Day 42, placebo.
  Interventions: Biological: Trivalent inactivated influenza vaccine; Biological: Inactivated H1N1 Vaccine; Drug: Placebo
- Group 4: TIV+placebo; H1N1+placebo; H1N1 (Experimental): 200 subjects (100 ages 18-64 years and 100 aged greater than or equal to 65 years) to receive: Day 0, trivalent influenza vaccine (TIV) + placebo; Day 21, 15 mcg H1N1 Vaccine + placebo; and Day 42, 15 mcg H1N1 vaccine.
  Interventions: Biological: Trivalent inactivated influenza vaccine; Biological: Inactivated H1N1 Vaccine; Drug: Placebo

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Licensed trivalent influenza vaccine (TIV) administered as a single 0.5 mL intramuscular injection in the deltoid muscle.
Biological: Inactivated H1N1 Vaccine — Two doses of inactivated influenza H1N1 vaccine, 15 mcg per dose, administered as a single 0.5 milliliters (mL) intramuscular injection in the deltoid muscle.
Drug: Placebo — Normal saline (placebo control) administered as a single 0.5 mL intramuscular injection in the deltoid muscle.

SUMMARY:
The purpose of this study is to assess the safety and immune response (body's defense against disease) to an experimental H1N1 influenza vaccine against the 2009 H1N1 virus. This study will help determine how the H1N1 flu shot should be given with the seasonal flu shot to make it most effective. Participants will include up to 850 healthy adults, ages 18 and older. Participants will receive 2 H1N1 vaccines in addition to placebo (inactive substance) and the seasonal flu shot over 3 study visits about 21 days apart. Study procedures include: medical history, physical exam, maintaining a memory aid, and blood sample collection. Participants will be involved in the study for about 8 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. Adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. If the novel influenza H1N1 2009 virus continues to circulate, it is possible that it will co-circulate with the non-pandemic seasonal influenza strains. In this situation, it might be beneficial to co-administer an H1N1 vaccine concurrent with the seasonal inactivated influenza vaccine. This protocol explores if vaccination with the 2009-2010 licensed seasonal trivalent influenza vaccine (TIV) has an effect on antibody response to the novel influenza H1N1 2009 virus and examines if receiving the H1N1 vaccine either concurrent with, prior to, or following the seasonal influenza vaccine affects the antibody response to the seasonal influenza vaccine. This is a randomized, double-blinded, Phase II study in up to 850 healthy males and non-pregnant females, aged 18 and older. The study investigates the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine when given concurrent with or sequentially with (before or after) TIV. The primary safety objective is to assess the safety of the unadjuvanted, inactivated H1N1 influenza vaccine when administered either concurrent with, prior to, or following licensed seasonal influenza vaccination. The primary immunogenicity objective is to assess the effect of TIV on antibody response to unadjuvanted, inactivated influenza H1N1 vaccine as assessed by hemagglutination inhibition assay (HAI), stratified by age of recipient. The secondary objective is immunogenicity, to assess the effect of H1N1 vaccine administration on antibody response to TIV as assessed by HAI, stratified by age of recipient. Subjects will be randomized into 4 groups, stratified by age (200 subjects per group with 100 subjects per age stratum, 18-64 or greater than or equal to 65 years of age). Group 1 will receive two 15 microgram (mcg) doses of H1N1 vaccine at Days 0 and 21 followed by TIV on Day 42. Group 2 will receive two 15 mcg doses of H1N1 vaccine of which the first dose is administered concurrently with TIV. Group 3 will receive two 15 mcg doses of H1N1 vaccine of which the second dose is administered concurrently with TIV. Group 4 will receive TIV administered on Day 0 followed by two 15 mcg doses of H1N1 vaccine on Days 21 and 42. In order to maintain the blind, subjects will also receive a placebo (normal saline) so that two products will be administered at both Days 0 and 21, and one product will be administered at Day 42 for all groups. Following immunization, safety will be measured by assessment of adverse events for 21 days following the last vaccination (Day 42 for those who do not receive the second dose), serious adverse events and new-onset chronic medical conditions for 8 months post the first vaccination (Day 222), and reactogenicity to the vaccines for 8 days following each vaccination (Day 0-7). Immunogenicity testing will include HAI

ELIGIBILITY:
Inclusion Criteria:

* Are males or non-pregnant females age 18 and older, inclusive.
* Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
* Are in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal and chicken protein).
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination (if female of childbearing potential), or women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 micrograms (mcg)/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during the study period (prior to Day 180 after the third vaccination).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the last vaccination.
* Has received a licensed 2009-2010 seasonal influenza vaccine.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have a history of severe reactions following previous immunization with influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 3 days prior to vaccination.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in a novel influenza H1N1 2009 vaccine study in the past two years or have a history of novel influenza H1N1 2009 infection prior to enrollment.
* Have known active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Plan to travel outside of North America in the time between the first vaccination and 63 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Saint Louis University Hospital - Internal Medicine - Infectious Diseases, Allergy & Immunology, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and females recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 7AUG2009 and 28AUG2009.
Groups:
- Group 1: H1N1+Placebo; H1N1+Placebo; TIV; Group 4: TIV+Placebo; H1N1+Placebo; H1N1: Participants received 15 mcg H1N1 Vaccine + saline placebo on Day 0; 15 mcg H1N1 Vaccine + saline placebo on Day 21, and Trivalent Influenza Vaccine (TIV) on Day 42
- Group 2: H1N1+TIV; H1N1+Placebo; Placebo: Participants received 15 mcg H1N1 Vaccine + Trivalent Influenza Vaccine (TIV) on Day 0; 15 mcg H1N1 Vaccine + saline placebo on Day 21, and saline placebo on Day 42
- Group 3: H1N1+Placebo; H1N1+TIV; Placebo: Participants received 15 mcg H1N1 Vaccine + saline placebo on Day 0; 15 mcg H1N1 Vaccine + Trivalent Influenza Vaccine (TIV) on Day 21, and saline placebo on Day 42
Period: Overall Study
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Started | 202 | 200 | 203 | 200
Completed | 200 | 198 | 197 | 198
Not Completed | 2 | 2 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1 | Total
Number analyzed (Participants) | 202 | 200 | 203 | 200 | 805
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 101 | 103 | 102 | 102 | 408
  >=65 years | 101 | 97 | 101 | 98 | 397
Age Continuous [Mean (Standard Deviation); unit: years] | 59.2 (16.2) | 58.4 (16.7) | 58.5 (16.6) | 59.1 (15.3) | 58.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 118 | 104 | 123 | 444
  Male | 103 | 82 | 99 | 77 | 361
Region of Enrollment [Number; unit: participants]
  United States | 202 | 200 | 203 | 200 | 805

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. For Group 4, this timepoint is Study Day 42, all others it is Study Day 21. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint, both within 4 days of the window, are included. Seven participants were excluded due to eligibility deviations, vaccine administration error or other protocol deviations. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 98 | 101 | 99 | 94
Participants | 90 | 87 | 91 | 82

2. Primary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 1
Time Frame: Day 21 after first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint, both within 4 days of the window, are included. One participant was excluded due to receipt of a non-study vaccine. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 101 | 97 | 101 | 95
Participants | 81 | 79 | 88 | 75

3. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; may have jeopardized the participant or required intervention to prevent one of these outcomes; or was described as Guillain-Barré Syndrome. Association to vaccination was determined by a study clinician licensed to make medical diagnoses.
Time Frame: Day 0 through Day 180 after the last vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 200 | 203 | 200
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post first H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more. Day 21 post first H1N1 vaccination is Study Day 42 for Group 4, and is Study Day 21 for all other groups.
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 98 | 101 | 99 | 94
Participants | 84 | 83 | 89 | 78

5. Secondary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: Blood was collected from participants for testing in the HAI assay against each strain in the 2009-2010 trivalent influenza vaccine. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 63 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 63 titer was an increase by 4-fold or more.
Time Frame: Day 63
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Eight participants were excluded due to eligibility deviations, vaccine administration error or other protocol deviations. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 91 | 89 | 88 | 90
Participants
  TIV H1 antigen | 46 | 40 | 38 | 39
  TIV H3 antigen | 52 | 48 | 46 | 47
  TIV B antigen | 34 | 31 | 36 | 39

6. Secondary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: as for outcome 5
Time Frame: Day 63
Population: Participants who received all vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Three participants were excluded due to receipt of non-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 92 | 87 | 90 | 91
Participants
  TIV H1 antigen | 66 | 62 | 53 | 57
  TIV H3 antigen | 37 | 27 | 34 | 31
  TIV B antigen | 14 | 14 | 20 | 18

7. Secondary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more. Day 21 post second H1N1 vaccination is Study Day 63 for Group 4, and is Study Day 42 for all other groups.
Time Frame: Day 0 prior to vaccination and 21 days after the second H1N1 vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Eight participants were excluded due to eligibility deviations, vaccine administration error or other protocol deviations. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 94 | 92 | 90 | 90
Participants | 85 | 77 | 85 | 75

8. Secondary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 7
Time Frame: Day 0 prior to vaccination and 21 days after the second H1N1 vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Three participants were excluded due to receipt of non-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 96 | 92 | 93 | 91
Participants | 80 | 73 | 72 | 65

9. Primary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 4
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint are included. One participant was excluded due to receipt of a non-study vaccine. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 101 | 97 | 101 | 95
Participants | 78 | 72 | 78 | 68

10. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, and nausea for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 200 | 203 | 200
Participants
  Feverishness | 12 | 12 | 7 | 13
  Malaise | 30 | 41 | 27 | 33
  Myalgia | 23 | 24 | 16 | 23
  Headache | 43 | 44 | 35 | 44
  Nausea | 12 | 11 | 11 | 12

11. Secondary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: Blood was collected from participants 21 days after the last vaccination for testing in the HAI assay against each strain in the 2009-2010 trivalent influenza vaccine. Each sample was tested according to standard operating procedures. A participant is counted if the value at the Day 63 timepoint was 1:40 or greater.
Time Frame: Day 63
Population: Participants who received all scheduled vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Eight participants were excluded due to eligibility deviations, vaccine administration error or other protocol deviations. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 91 | 89 | 88 | 90
Participants
  TIV H1 antigen | 79 | 77 | 78 | 81
  TIV H3 antigen | 84 | 80 | 77 | 84
  TIV B antigen | 81 | 75 | 78 | 81

12. Secondary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the Virus Strains in the 2009-2010 Trivalent Influenza Vaccine (TIV) 21 Days Following the Last Vaccination
Description: as for outcome 11
Time Frame: Day 63
Population: Participants who received all scheduled vaccinations and from whom blood was collected at the timepoint, all within 4 days of the window, are included. Three participants were excluded due to receipt of non-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 92 | 87 | 90 | 91
Participants
  TIV H1 antigen | 85 | 82 | 81 | 87
  TIV H3 antigen | 86 | 80 | 83 | 77
  TIV B antigen | 71 | 69 | 68 | 62

13. Secondary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. For Group 4, this timepoint is Study Day 63, all others it is Study Day 42. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after second H1N1 vaccination
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 94 | 92 | 90 | 90
Participants | 89 | 82 | 87 | 80

14. Secondary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 13
Time Frame: Day 21 after second H1N1 vaccination
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 96 | 92 | 93 | 91
Participants | 83 | 78 | 81 | 71

15. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 10
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 193 | 190 | 189 | 192
Participants
  Feverishness | 14 | 8 | 12 | 10
  Malaise | 29 | 29 | 35 | 23
  Myalgia | 18 | 14 | 19 | 14
  Headache | 28 | 26 | 29 | 21
  Nausea | 6 | 6 | 4 | 8

16. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the Third Vaccination
Description: as for outcome 10
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: Participants who received the third vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 190 | 185 | 183 | 188
Participants
  Feverishness | 6 | 8 | 5 | 5
  Malaise | 17 | 15 | 18 | 14
  Myalgia | 10 | 12 | 11 | 6
  Headache | 16 | 19 | 17 | 15
  Nausea | 4 | 5 | 5 | 7

17. Primary Outcome: Number of Participants Reporting Fever After the First Vaccination
Description: Participants were provided a thermometer and a memory aid to record daily oral temperatures for 8 days (Day 0-7) after vaccination. Participants are counted as experiencing fever if they reported oral temperatures of 38 degrees Celsius or higher on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: Participants who received the first vaccination and reported oral temperatures during the time period are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 200 | 202 | 200
Participants | 0 | 1 | 0 | 0

18. Primary Outcome: Number of Participants Reporting Fever After the Second Vaccination
Description: as for outcome 17
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: Participants who received the second vaccination and reported oral temperatures during the time period are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 193 | 190 | 188 | 192
Participants | 0 | 2 | 0 | 3

19. Primary Outcome: Number of Participants Reporting Fever After the Third Vaccination
Description: as for outcome 17
Time Frame: Within 8 days (Day 0-7) post third vaccination
Population: Participants who received the third vaccination and reported oral temperatures during the time period are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 190 | 184 | 183 | 188
Participants | 0 | 0 | 1 | 0

20. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the First H1N1 Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days. First H1N1 vaccination was given on Study Day 0 for Groups 1, 2 and 3, and on Study Day 21 for Group 4.
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: Participants who received the first H1N1 vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 200 | 203 | 192
Participants
  Pain | 26 | 32 | 26 | 11
  Tenderness | 45 | 46 | 47 | 29
  Swelling | 18 | 14 | 16 | 20

21. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the Second H1N1 Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days. Second H1N1 vaccination was given on Study Day 21 for Groups 1, 2 and 3, and on Study Day 42 for Group 4.
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: Participants who received the second H1N1 vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 194 | 190 | 189 | 188
Participants
  Pain | 28 | 22 | 30 | 19
  Tenderness | 51 | 44 | 58 | 37
  Swelling | 28 | 17 | 20 | 25

22. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the TIV Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days. The TIV vaccination was given on Study Day 42 for Group 1, Study Day 0 for Groups 2 and 4, and on Study Day 21 for Group 3.
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: Participants who received the TIV vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 190 | 200 | 189 | 200
Participants
  Pain | 32 | 57 | 46 | 48
  Tenderness | 71 | 93 | 80 | 84
  Swelling | 27 | 27 | 22 | 28

23. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the First Placebo Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days. The first placebo vaccination was given on Study Day 0 for Groups 1, 3 and 4, and on Study Day 21 for Group 2.
Time Frame: Within 8 days (Day 0-7) post first placebo vaccination
Population: Participants who received the first placebo vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 190 | 203 | 200
Participants
  Pain | 12 | 14 | 13 | 11
  Tenderness | 21 | 14 | 21 | 21
  Swelling | 12 | 18 | 12 | 14

24. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the Second Placebo Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days. The second placebo vaccination was given on Study Day 21 for Groups 1 and 4, on Study Day 42 for Groups 2 and 3.
Time Frame: Within 8 days (Day 0-7) post second placebo vaccination
Population: Participants who received the second placebo vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 194 | 185 | 183 | 192
Participants
  Pain | 11 | 9 | 5 | 8
  Tenderness | 15 | 7 | 9 | 17
  Swelling | 25 | 13 | 14 | 13

25. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the First H1N1 Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first H1N1 vaccination
Population: Participants who received the first H1N1 vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 200 | 203 | 192
Participants
  Redness | 32 | 33 | 27 | 31
  Swelling | 19 | 16 | 19 | 21

26. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the Second H1N1 Vaccination
Description: as for outcome 25
Time Frame: Within 8 days (Day 0-7) post second H1N1 vaccination
Population: Participants who received the second H1N1 vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 194 | 190 | 189 | 188
Participants
  Redness | 29 | 27 | 29 | 35
  Swelling | 29 | 18 | 19 | 27

27. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the TIV Vaccination
Description: as for outcome 25
Time Frame: Within 8 days (Day 0-7) post TIV vaccination
Population: Participants who received the TIV vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 190 | 200 | 189 | 200
Participants
  Redness | 31 | 40 | 30 | 37
  Swelling | 28 | 27 | 21 | 28

28. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the First Placebo Vaccination
Description: as for outcome 25
Time Frame: Within 8 days (Day 0-7) post first placebo vaccination
Population: Participants who received the first placebo vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 202 | 190 | 203 | 200
Participants
  Redness | 34 | 19 | 21 | 37
  Swelling | 12 | 20 | 12 | 28

29. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the Second Placebo Vaccination
Description: as for outcome 25
Time Frame: Within 8 days (Day 0-7) post second placebo vaccination
Population: Participants who received the second placebo vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Number analyzed (Participants) | 194 | 185 | 183 | 192
Participants
  Redness | 30 | 25 | 26 | 30
  Swelling | 27 | 17 | 14 | 14

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | Group 1: H1N1+Placebo; H1N1+Placebo; TIV | Group 2: H1N1+TIV; H1N1+Placebo; Placebo | Group 3: H1N1+Placebo; H1N1+TIV; Placebo | Group 4: TIV+Placebo; H1N1+Placebo; H1N1
Serious Adverse Events (participants affected / at risk) | 5/202 | 7/200 | 12/203 | 13/200
Other Adverse Events (participants affected / at risk) | 167/202 | 170/200 | 169/203 | 175/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: H1N1+Placebo; H1N1+Placebo; TIV (N=202) | Group 2: H1N1+TIV; H1N1+Placebo; Placebo (N=200) | Group 3: H1N1+Placebo; H1N1+TIV; Placebo (N=203) | Group 4: TIV+Placebo; H1N1+Placebo; H1N1 (N=200)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypervitaminosis A (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: H1N1+Placebo; H1N1+Placebo; TIV (N=202) | Group 2: H1N1+TIV; H1N1+Placebo; Placebo (N=200) | Group 3: H1N1+Placebo; H1N1+TIV; Placebo (N=203) | Group 4: TIV+Placebo; H1N1+Placebo; H1N1 (N=200)
Injection site haematoma (General disorders) | 18 (18) | 30 (35) | 20 (26) | 18 (20)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 12 (12) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6) | 4 (4) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 18 (18) | 23 (23) | 18 (19)
Feeling hot (General disorders) | 26 (32) | 24 (28) | 20 (24) | 24 (28)
Malaise (General disorders) | 59 (76) | 61 (85) | 57 (80) | 55 (70)
Myalgia (Musculoskeletal and connective tissue disorders) | 42 (51) | 40 (50) | 39 (46) | 37 (43)
Headache (Nervous system disorders) | 64 (87) | 62 (89) | 60 (81) | 60 (80)
Nausea (Gastrointestinal disorders) | 18 (22) | 21 (22) | 16 (20) | 22 (27)
Injection site pain (General disorders) | 66 (97) | 87 (109) | 72 (91) | 67 (89)
Tenderness (General disorders) | 98 (184) | 115 (159) | 111 (162) | 109 (166) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 73 (115) | 67 (107) | 71 (97) | 75 (118)
Injection site swelling (functional grading) (General disorders) | 57 (88) | 56 (73) | 50 (67) | 59 (84) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 61 (93) | 59 (81) | 52 (69) | 61 (89) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less